CLINICAL TRIAL: NCT07139834
Title: Examining the Effects of Escitalopram and Memantine on Pattern Separation in Major Depressive Disorder
Brief Title: Pattern Separation in Major Depressive Disorder
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey Miller (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Miller, Research Scientist, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 00081503
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression; Major depressive disorder; MDD; Pattern separation; Memantine
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Selective Serotonin Reuptake Inhibitors; Escitalopram; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study coordinator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SSRI + Memantine (Experimental)
  Interventions: Drug: SSRI (escitalopram or sertraline); Drug: Extended-Release Memantine
- SSRI + Placebo (Placebo Comparator)
  Interventions: Drug: SSRI (escitalopram or sertraline); Drug: Placebo

INTERVENTIONS:
Drug: SSRI (escitalopram or sertraline) — 11 weeks of open-label treatment with an SSRI, of which the last 6 weeks are augmented with memantine vs placebo. Primary SSRI for the study is escitalopram. In cases of prior intolerance or non-response to escitalopram, individuals will be treated with sertraline instead of escitalopram.
Drug: Extended-Release Memantine — 6 weeks of treatment with extended-release memantine as augmentation to ongoing escitalopram treatment
  Arms: SSRI + Memantine
Drug: Placebo — 6 weeks of treatment with placebo as augmentation to ongoing escitalopram treatment
  Arms: SSRI + Placebo

SUMMARY:
This study seeks to examine the effects of treatment with a selective serotonin reuptake inhibitor (SSRI), escitalopram, a first-line treatment for depression, in combination with placebo or with extended-release memantine, on neuropsychological function, regional brain activity assessed by functional magnetic resonance imaging, and depressive symptoms, in participants with Major Depressive Disorder. Escitalopram is administered in an open-label fashion in this study; extended release memantine is administered in a double-blind, randomized, placebo-controlled manner.

DETAILED DESCRIPTION:
Pattern separation is the process of separating overlapping sensory information, contexts, or experiences into distinct neural representations. In humans, deficits in pattern separation are believed to underlie overgeneralization seen in depression and post-traumatic stress disorder (PTSD). Cross-sectional data support the effects of SSRI medications on pattern separation. Specifically, a recent paper demonstrated patients with depression who responded to SSRI medication had improved pattern separation performance (mnemonic discrimination) of emotionally neutral stimuli than SSRI non-responders, and that the findings were reversed with respect to emotionally negative stimuli (Phillips et al., 2023). These data are consistent with the negative cognitive bias in depression (Beevers et al., 2019), and provide indirect evidence of SSRI effects on pattern separation in humans. However, there is a dearth of longitudinal, within-subject analyses of SSRI effects on pattern separation performance, and associated neural activity quantified by BOLD signal from fMRI.

In the current study, we seek to examine the individual effect of SSRI treatment (in combination with placebo) as compared to the combined effect of treatment with SSRI and memantine, an NMDA-antagonist, on pattern separation, both in terms of behavioral performance and activity in the dentate gyrus as assessed by fMRI, and on depression severity. We propose to study individuals with major depressive disorder in a current major depressive episode who are currently unmedicated, who will undergo baseline medical and psychiatric assessment and fMRI scanning, followed by standardized treatment with escitalopram combined with either placebo or memantine in the context of a double-blind, placebo-controlled, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Current diagnosis of MDD without psychotic features assessed within three weeks of study enrollment
* 17-item Hamilton Depression Rating Scale score ≥17 assessed within 3 weeks of study enrollment
* Using an effective form of contraception at study enrollment and agrees to continue throughout study participation for individuals of child-bearing potential
* Capacity to provide informed consent
* Proficient in English
* Willing to provide emergency contact

Exclusion Criteria:

* Currently taking an antidepressant medication at study enrollment
* Pregnant or breastfeeding at time of enrollment
* Evidence of current unstable medical illness, including liver or renal impairment, or unstable cardiovascular or respiratory illness
* QTc interval greater than 500 ms
* Current genitourinary conditions that raise urine pH such as a) renal tubular acidosis or b) severe infection of the urinary tract.
* Clinically significant neurological conditions, including a) history of stroke, b) previous head injury with evidence of cognitive impairment, c) history of malignancy or d) history of seizure disorder. (headache, migraines, pain disorders, and other conditions not exclusionary)
* Lifetime diagnosis of a) bipolar disorder, b) psychotic disorder, or c) dementia
* Current active suicidal ideation
* Current substance use disorder other than tobacco use disorder
* Current or recent (past 6 months) treatment with antipsychotics; current or recent (past 1 month) treatment with benzodiazepines; current use of prescribed stimulant medication; current use of other NMDA antagonists (amantadine, ketamine, dextromethorphan)
* Current use of disulfiram with oral concentrate, MAOIs (including linezolid or IV methylene blue), or pimozide
* History of hypersensitivity or allergic reaction to a) memantine hydrochloride or any of its components/excipients, b) citalopram, escitalopram, or any other component of the product, or c) sertraline or any other component of the product
* Concurrent or recent (past 6 months) participation in another clinical trial for mental illness involving an investigational product or device
* Lack of response to or intolerable side-effects from trials of two or more selective serotonin reuptake inhibitors of adequate dose and duration at study enrollment
* Electroconvulsive therapy (ECT) in the past 6 months
* Any condition or material in the body that is a contraindication for MRI procedures
* Weight that exceeds 300 lbs or inability to fit into MRI scanner
* MST LDI score greater than 0.5

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Pattern Separation Performance | At baseline (week 0) and after completing the medication trial (week 11)
  Participants will complete a pattern separation task

SECONDARY OUTCOMES:
Depression Severity | At screening, baseline (week 0) and after completing the medication trial (week 11)
  Depression severity will be assessed using the Montgomery-Asberg Depression Rating Scale (MADRS)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Miller, MD, Principal Investigator — New York State Psychiatric Institute (NYSPI)
Locations (1):
- New York State Psychiatric Institute (NYSPI), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from this study may be shared with other investigators, including neuroimaging, neurocognitive, diagnostic, demographic, and clinical ratings data.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information will be made available within one year following the conclusion of study recruitment, with no specified end point.
Access Criteria: Sharing of the IPD described above with investigators outside the study team will occur through institutionally approved mechanisms that may require a data use agreement. Requests for sharing of IPD can be made to the study's principal investigator, who will confirm that all institutional requirements are met prior to data sharing.

REFERENCES:
- [Background] Beevers CG, Mullarkey MC, Dainer-Best J, Stewart RA, Labrada J, Allen JJB, McGeary JE, Shumake J. Association between negative cognitive bias and depression: A symptom-level approach. J Abnorm Psychol. 2019 Apr;128(3):212-227. doi: 10.1037/abn0000405. Epub 2019 Jan 17. PMID 30652884
- [Background] Phillips TO, Castro M, Vas RK, Ferguson LA, Harikumar A, Leal SL. Perceived antidepressant efficacy associated with reduced negative and enhanced neutral mnemonic discrimination. Front Hum Neurosci. 2023 Aug 28;17:1225836. doi: 10.3389/fnhum.2023.1225836. eCollection 2023. PMID 37701502